CLINICAL TRIAL: NCT07317063
Title: An Open-label, Single-center Trial Evaluating the Safety, Tolerability, and Pharmacokinetics of a Single Dose of GRT6019, Including Food Effect, in Healthy Male Participants
Brief Title: A Trial to Investigate Safety and Pharmacokinetics of GRT6019, Including Food Effect, in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Grünenthal GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP6019-10
Record Dates: First submitted 2025-12-19; First posted 2026-01-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Duchenne Muscular Dystrophy (DMD)
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Fed State
  Interventions: Drug: GRT6019
- Cohort 2 (Experimental): Fasted State
  Interventions: Drug: GRT6019

INTERVENTIONS:
Drug: GRT6019 — Single Dose

SUMMARY:
The purpose of this trial is to evaluate the safety, tolerability, and Pharmacokinetics (PK) of a single oral dose of GRT6019 in healthy male participants, including food effect.

This is an open-label, single-dose, single-center Phase I trial with healthy male participants. The trial will consist of 2 cohorts with a total duration of approximately 7 weeks, including a 28-day Screening Period.

The participants will receive a single dose of GRT6019 administered on Day 1 and will remain at the clinic for 7 additional days.

Following the in-house stay, there will be 2 Follow-up Visits up until Day 23, with 3 clinic visits scheduled

DETAILED DESCRIPTION:
Cohort 1 and Cohort 2 will be dosed in parallel:

* Cohort 1 (n = 9): single dose of GRT6019 in participants in a fed state
* Cohort 2 (n = 9): single dose of GRT6019 in participants in a fasted state

ELIGIBILITY:
Main inclusion Criteria:

1. The participant must be able to give signed informed consent, including compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Participants must sign the ICF before any trial-related assessments.
3. The participant is in good health as determined by the medical history, physical examination, 12-lead Electrocardiogram (ECG), vital signs (heart rate [HR], respiratory rate [RR], systolic and diastolic blood pressure [BP]), body temperature, and clinical laboratory parameters (clinical chemistry, hematology, coagulation, and urinalysis) without clinically relevant (per investigator judgement) deviations from reference ranges unless further specified in the exclusion criteria.

Main exclusion Criteria:

1. Any disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding that contraindicates the use of an investigational drug, comparator, rescue medication, or any ingredients therein, or may affect the interpretation of the results, or may render the patient at high risk from treatment complications/ participation in the study unsafe.
2. Major surgical procedure, within 3 months prior to ICF signing, or anticipation of need for a major surgical procedure during the trial.
3. Clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, or immunological disorder(s) as determined by the investigator.
4. Any medication, including herbal remedies or over-the-counter medication within 2 weeks before screening into this trial and anticipated use during the trial.
5. Concurrent enrollment in another clinical trial unless it is an observational (non-interventional) clinical trial or during the Follow-up Period of an interventional trial.
6. Recent participation in another clinical trial with an IMP administered within 30 days before Day 1 OR within 5 times the elimination half-life of the IMP, whichever is longer.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2025-11-21 (Actual); Primary Completion 2026-01-06 (Actual); Study Completion 2026-01-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events | Through study completion, an average of 7 Weeks
  Assessment of safety and tolerability of GRT6019 after a single oral dose
Number of participants with serious Adverse Events | Through study completion, an average of 7 Weeks
  Assessment of safety and tolerability of GRT6019 after a single oral dose
Number of participants with Adverse Events leading to discontinuation | Through study completion, an average of 7 Weeks
  Assessment of safety and tolerability of GRT6019 after a single oral dose
Number of participants with Adverse Events related with GRT6019 | Through study completion, an average of 7 Weeks
  Assessment of safety and tolerability of GRT6019 after a single oral dose

SECONDARY OUTCOMES:
Area under the concentration-time curve from pre-dose (time 0) to the time of the last quantifiable concentration (AUC0-t) | From pre-dose (at -2 hours to -5 minutes ) to 528 hours post-dose.
  The total amount of the study drug in the blood from the time it is taken until the last time a measurable level of the drug is found.
  Assessment of the PK of GRT6019 following a single dose under fasted and fed conditions.
Area under the concentration-time curve from pre-dose (time 0) extrapolated to infinite time (AUC0-inf ) | From pre-dose (at -2 hours to -5 minutes ) to 528 hours post-dose.
  The total amount of the study drug in the blood from the time it is taken until it has completely left the body.
  Assessment of the PK of GRT6019 following a single dose under fasted and fed conditions.
Maximum plasma concentration (Cmax) | From pre-dose (at -2 hours to -5 minutes ) to 528 hours post-dose.
  The maximum amount of the study drug measured in the blood after taking the dose.
  Assessment of the PK of GRT6019 following a single dose under fasted and fed conditions.
Time of maximum plasma concentration (Tmax) | From pre-dose (at -2 hours to -5 minutes ) to 528 hours post-dose.
  The time it takes to reach the highest concentration of the study drug in the blood after dosing.
  Assessment of the PK of GRT6019 following a single dose under fasted and fed conditions.
Lag-time observed from dosing to the time point prior to that of the first quantifiable plasma concentration (Tlag). Assessment of the PK of GRT6019 following a single oral dose of the pediatric formulation under fasted and fed conditions. | From pre-dose (at -2 hours to -5 minutes ) to 528 hours post-dose.
  The time between when the study drug is taken and when it first becomes measurable in the blood.
  Assessment of the PK of GRT6019 following a single dose under fasted and fed conditions.
Terminal elimination half life (T₁/₂) | From pre-dose (at -2 hours to -5 minutes ) to 528 hours post-dose.
  The time it takes for the amount of study drug in the blood to reduce by half after reaching its peak level.
  Assessment of the PK of GRT6019 following a single dose under fasted and fed conditions.
Total body oral clearance (CL/F) | From pre-dose (at -2 hours to -5 minutes ) to 528 hours post-dose.
  The amount of blood completely cleared of thestudy drug (and metabolite) per unit of time, taking into account how much of the drug is absorbed into the body.
  Assessment of the PK of GRT6019 following a single dose under fasted and fed conditions.
Apparent volume of distribution (V/F) | From pre-dose (at -2 hours to -5 minutes ) to 528 hours post-dose.
  An estimate of how widely the study drug spreads through the body's tissues after it is absorbed.
  Assessment of the PK of GRT6019 following a single dose under fasted and fed conditions.
Ratio of the geometric mean of AUC0-t | From pre-dose (at -2 hours to -5 minutes ) to 528 hours post-dose.
  Assessment of the effect of food (fed and fasted state) on the PK of GRT6019 following a single dose.
Ratio of the geometric mean of AUC0-inf | From pre-dose (at -2 hours to -5 minutes ) to 528 hours post-dose.
  Assessment of the effect of food (fed and fasted state) on the PK of GRT6019 following a single dose.
Ratio of the geometric mean of Cmax | From pre-dose (at -2 hours to -5 minutes ) to 528 hours post-dose.
  Assessment of the effect of food (fed and fasted state) on the PK of GRT6019 following a single dose.

CONTACTS AND LOCATIONS:
Locations (1):
- Biotrial, Inc, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No